CLINICAL TRIAL: NCT05532592
Title: Investigation on the Hesitancy of COVID-19 Vaccination Among Liver Transplant Recipients in China
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yongbing Qian, associate chief physician, RenJi Hospital
Other Study IDs: KY2022-138-B
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Vaccine Hesitancy
Keywords: COVID-19; vaccine; vaccine hesitancy; liver transplant recipients; China
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no hesitancy group (NHG): Participants who got vaccine after transplantation or were willing to be vaccinated.
  Interventions: Other: Perceptions and attitudes towards COVID-19 and COVID-19 vaccine
- hesitancy group (HG): Participants who were uncertain or refused to be vaccinated.
  Interventions: Other: Perceptions and attitudes towards COVID-19 and COVID-19 vaccine

INTERVENTIONS:
Other: Perceptions and attitudes towards COVID-19 and COVID-19 vaccine — Attitude towards COVID-19; Knowledge about COVID-19 vaccine

SUMMARY:
On WeChat platform, through a point-to-point connection, and carry on the questionnaire survey to collect information of liver transplant recipients followed-up by the department of Liver Surgery, Renji Hospital Shanghai Jiao Tong University. Patients meeting inclusion and exclusion criteria will be selected. Conduct statistical analysis to describe the incidence of adverse reactions related to COVID-19 vaccine after liver transplantation, and to compare and evaluate the factors leading to COVID-19 vaccine hesitancy.

DETAILED DESCRIPTION:
On WeChat platform, through a point-to-point connection, and carry on the questionnaire survey to collect information of liver transplant recipients followed-up by the department of Liver Surgery, Renji Hospital Shanghai Jiao Tong University. Questionnaire items including demographic characteristics, understanding of COVID-19, attitude toward COVID-19 vaccine. Patients meeting inclusion and exclusion criteria will be selected. Conduct statistical analysis to describe the incidence of adverse reactions related to COVID-19 vaccine after liver transplantation, and to compare and evaluate the factors leading to COVID-19 vaccine hesitancy.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. recipients after liver transplantation surgery

Exclusion Criteria:

1. Incomplete data (missing questionnaire information), such as lack of age, gender, indication for transplantation, time after transplantation and other indicators
2. loss to follow-up
3. COVID-19 vaccination before liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of this study were adult recipients who were followed up after liver transplantation in the department of Liver Surgery, Renji Hospital Shanghai Jiao Tong University.
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with COVID-19 Vaccine Hesitancy | through study completion, an average of 1 year
  In the questionnaire, participants who expressed hesitancy or explicitly refused to receive the COVID-19 vaccine were considered vaccine hesitancy.

CONTACTS AND LOCATIONS:
Overall Officials: Yongbing Qian, Prof, Study Director — The department of Liver Surgery, Renji Hospital Shanghai Jiao Tong University.
Locations (1):
- The department of Liver Surgery, Renji Hospital Shanghai Jiao Tong University., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
This retrospective study involves the privacy of the participants. We need to keep it confidential and do not plan to share the data. If you want to know the relevant information, you can contact the principal person in charge of the study

REFERENCES:
- [Background] Azzi Y, Bartash R, Scalea J, Loarte-Campos P, Akalin E. COVID-19 and Solid Organ Transplantation: A Review Article. Transplantation. 2021 Jan 1;105(1):37-55. doi: 10.1097/TP.0000000000003523. PMID 33148977
- [Background] Stucchi RSB, Lopes MH, Kumar D, Manuel O. Vaccine Recommendations for Solid-Organ Transplant Recipients and Donors. Transplantation. 2018 Feb;102(2S Suppl 2):S72-S80. doi: 10.1097/TP.0000000000002012. No abstract available. PMID 29381581
- [Background] Russo FP, Piano S, Bruno R, Burra P, Puoti M, Masarone M, Montagnese S, Ponziani FR, Petta S, Aghemo A; Italian Association for the Study of the Liver. Italian association for the study of the liver position statement on SARS-CoV2 vaccination. Dig Liver Dis. 2021 Jun;53(6):677-681. doi: 10.1016/j.dld.2021.03.013. Epub 2021 Apr 30. PMID 33941488
- [Background] Cornberg M, Buti M, Eberhardt CS, Grossi PA, Shouval D. EASL position paper on the use of COVID-19 vaccines in patients with chronic liver diseases, hepatobiliary cancer and liver transplant recipients. J Hepatol. 2021 Apr;74(4):944-951. doi: 10.1016/j.jhep.2021.01.032. Epub 2021 Feb 6. PMID 33563499
- [Background] Fix OK, Blumberg EA, Chang KM, Chu J, Chung RT, Goacher EK, Hameed B, Kaul DR, Kulik LM, Kwok RM, McGuire BM, Mulligan DC, Price JC, Reau NS, Reddy KR, Reynolds A, Rosen HR, Russo MW, Schilsky ML, Verna EC, Ward JW, Fontana RJ; AASLD COVID-19 Vaccine Working Group. American Association for the Study of Liver Diseases Expert Panel Consensus Statement: Vaccines to Prevent Coronavirus Disease 2019 Infection in Patients With Liver Disease. Hepatology. 2021 Aug;74(2):1049-1064. doi: 10.1002/hep.31751. PMID 33577086
- [Background] Facciola A, Visalli G, Orlando A, Bertuccio MP, Spataro P, Squeri R, Picerno I, Di Pietro A. Vaccine hesitancy: An overview on parents' opinions about vaccination and possible reasons of vaccine refusal. J Public Health Res. 2019 Mar 11;8(1):1436. doi: 10.4081/jphr.2019.1436. eCollection 2019 Mar 11. PMID 30997357
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383
- [Background] Chen T, Li X, Li Q, Huang L, Cai Q, Wang Y, Jiang Y, Xu Q, Lv Q, Wang J. COVID-19 vaccination hesitancy and associated factors among solid organ transplant recipients in China. Hum Vaccin Immunother. 2021 Dec 2;17(12):4999-5006. doi: 10.1080/21645515.2021.1984133. Epub 2021 Sep 29. PMID 34586945
- [Background] Costantino A, Invernizzi F, Centorrino E, Vecchi M, Lampertico P, Donato MF. COVID-19 Vaccine Acceptance among Liver Transplant Recipients. Vaccines (Basel). 2021 Nov 11;9(11):1314. doi: 10.3390/vaccines9111314. PMID 34835245
- See also: World Health Organization (WHO). Draft landscape of COVID-19 candidate vaccines. 2021 June 15. — https://www.who.int/publications/m/item/draft-landscape-of-covid-19-candidate-vaccines